CLINICAL TRIAL: NCT00268437
Title: A Phase II Trial of Preoperative Radiation and Chemotherapy (Pemetrexed and Carboplatin) for Locally Advanced Esophageal Cancer
Brief Title: Radiation Therapy, Pemetrexed Disodium, and Carboplatin in Treating Patients With Locally Advanced Esophageal Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial closed early because, during an interim analysis, the primary endpoint fell short.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N044E; NCI-2012-02678 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000455635 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage III esophageal cancer; stage II esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; Pemetrexed; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed/Carboplatin (Experimental): Pemetrexed+Carboplatin+Radiation
  Interventions: Drug: carboplatin; Drug: Pemetrexed; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — carboplatin is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.
Drug: Pemetrexed — Pemetrexed is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy — Radiation therapy begins day 1 and continues for 5 ½ weeks (45 Gy in 22-25 fractions of 1.8 Gy to extended field; 50.4 Gy in 28 fractions within boost field).

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as pemetrexed disodium and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving radiation therapy together with pemetrexed disodium and carboplatin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with pemetrexed disodium and carboplatin works in treating patients with locally advanced esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathologic complete response rate of radiotherapy, pemetrexed disodium, and carboplatin when administered prior to esophagectomy in patients with locally advanced esophageal cancer.

Secondary

* Determine the activity, in terms of clinical response rate and adverse event profile of radiotherapy, pemetrexed disodium, and carboplatin when administered prior to esophagectomy.
* Determine the overall survival, time-to-progression, and time-to-treatment failure for patients receiving the above combined modality treatment.
* Determine the surgical outcome for all patients who undergo esophagectomy.
* Determine the time-to-disease recurrence and disease-free survival for patients who have a curative resection.
* Determine quality of life of patients treated with this regimen. OUTLINE: This is a multicenter study. Patients undergo radiotherapy once daily, 5 days a week, for 5 ½ weeks and concurrently receive pemetrexed disodium IV over 10 minutes and carboplatin IV over 30 minutes on days 1 and 22. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who are eligible will undergo esophagectomy between 4-12 weeks after completion of radiotherapy.

Quality of life is assessed at baseline, immediately prior to day 22 of chemotherapy, and within 2 weeks prior to surgery.

After completion of study treatment, patients are followed periodically for approximately 4 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal (GE) junction

  * No T1-2, N0, M0 disease
  * No palpable or biopsy-proven involvement of supraclavicular nodes or radiographically involved supraclavicular nodes (> 1.5 cm in greatest dimension) for lesions in mid-thoracic, distal thoracic, or GE junction

    + Supraclavicular node involvement allowed provided there are upper thoracic esophagus primary lesions
  * Patients with involvement of celiac nodes (stations 15-20) are eligible if the primary lesion is mid-thoracic, distal esophagus, or GE junction
  * No evidence of distant metastases
* Tumor must be considered surgically resectable

  - Patients with T4, N0 tumors that are potentially resectable are eligible
* No clinically relevant pleural or peritoneal effusion that is not amenable to drainage

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥1,500/mm^3
* Platelet count ≥100,000/mm^3
* Hemoglobin ≥10 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine clearance ≥ 45 mL/min
* No New York Heart Association class III or IV congestive heart failure
* Pregnant or nursing women are ineligible
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other severe underlying disease that would preclude study entry
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ
* No prior sensitivity or allergic reaction to pemetrexed disodium or carboplatin
* Able to swallow pills

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for esophageal cancer
* No prior radiotherapy field that overlapped the anticipated fields of study radiotherapy
* No prior radiotherapy to > 30% of the marrow cavity
* Patients taking nonsteroidal anti-inflammatory drugs (NSAIDs) must be able to discontinue use 2 days prior, during, and 2 days after pemetrexed disodium administration (5 days prior for long-life NSAIDs)
* Patients must not have been receiving cyclooxygenase-2 inhibitors at study entry and while receiving protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (90):
- United States (90):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jatoi A, Soori G, Foster NR, Hiatt BK, Knost JA, Fitch TR, Callister MD, Nichols FC 3rd, Husted TM, Alberts SR. Phase II study of preoperative pemetrexed, carboplatin, and radiation followed by surgery for locally advanced esophageal cancer and gastroesophageal junction tumors. J Thorac Oncol. 2010 Dec;5(12):1994-8. doi: 10.1097/JTO.0b013e3181fb5c3e. PMID 20975604
- [Result] Katipamula R, Jatoi A, Foster NR, Nichols F, Rubin J, Callister M, Gunderson L, Alberts S. Pemetrexed, Carboplatin, and Concomitant Radiation followed by Surgery for Locally Advanced Esophageal Cancer: Results of a Planned Interim Toxicity Analysis of North Central Cancer Treatment Group Study N044E. Clin Med Oncol. 2008;2:223-5. doi: 10.4137/cmo.s444. Epub 2008 Apr 1. PMID 21892283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial closed early because, during an interim analysis, the primary endpoint fell short. However, 26 eligible patients were accrued. Due to early closure not all the endpoints were analyzed.
Groups:
- Pemetrexed/Carboplatin: Pemetrexed+Carboplatin+Radiation carboplatin: carboplatin is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.
  Pemetrexed: Pemetrexed is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.
  Radiation therapy: Radiation therapy begins day 1 and continues for 5 ½ weeks (45 Gy in 22-25 fractions of 1.8 Gy to extended field; 50.4 Gy in 28 fractions within boost field).
  Conventional surgery
Period: Overall Study
Arm/Group | Pemetrexed/Carboplatin
Started | 27
Completed | 26
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed/Carboplatin: Pemetrexed+Carboplatin+Radiation>
  > carboplatin: carboplatin is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.>
  > Pemetrexed: Pemetrexed is to be given on days 1 and 22 of the 5 ½ weeks of radiation treatment.>
  > conventional surgery>
  > neoadjuvant therapy>
  > radiation therapy: Radiation therapy begins day 1 and continues for 5 ½ weeks (45 Gy in 22-25 fractions of 1.8 Gy to extended field; 50.4 Gy in 28 fractions within boost field).
Arm/Group | Pemetrexed/Carboplatin
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 66 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: The proportion of pathologic complete responses will be estimated by the number of pathologic complete responses divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true pathologic complete response rate will be calculated. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for Measurable disease is defined as at least one lesion whose longest diameter can be accurately measured as ≥2.0 cm with conventional techniques or as ≥1.0 cm with spiral CT. Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung. However, CT is preferable.
Time Frame: Baseline to time of surgery (around 10 - 18 weeks post-baseline)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed/Carboplatin
Number analyzed (Participants) | 26
percentage of participants | 23 [9 to 44]

2. Secondary Outcome: Overall Survival
Description: Time from registration to death due to any cause.
Time Frame: From baseline to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed/Carboplatin
Number analyzed (Participants) | 26
months | 17.8 [12.2 to 30.7]

ADVERSE EVENTS:
Arm/Group | Pemetrexed/Carboplatin
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Carboplatin (N=27)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Carboplatin (N=27)
Hemoglobin decreased (Blood and lymphatic system disorders) | 25 (59)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 11 (15)
Dysphagia (Gastrointestinal disorders) | 20 (48)
Esophageal mucositis (Gastrointestinal disorders) | 7 (10)
Esophageal pain (Gastrointestinal disorders) | 11 (21)
Esophagitis (Gastrointestinal disorders) | 16 (30)
Nausea (Gastrointestinal disorders) | 19 (36)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 7 (9)
Vomiting (Gastrointestinal disorders) | 9 (12)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (12)
Endocarditis infective (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Small intestine infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Blood bilirubin increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 24 (43)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 23 (37)
Platelet count decreased (Investigations) | 23 (47)
Weight loss (Investigations) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (8)
Depression (Psychiatric disorders) | 5 (5)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (12)
Hypotension (Vascular disorders) | 7 (10)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes